CLINICAL TRIAL: NCT04656925
Title: Automated Reinforcement Management System (ARMS): Phase I Study
Brief Title: Automated Reinforcement Management System (ARMS)
Acronym: ARMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Sterling McPherson, Professor, Washington State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 18376
Record Dates: First submitted 2020-09-15; First posted 2020-12-07 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: A-B-A, or a return to baseline design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency management A-B-A (Experimental): All participants will be assigned a single arm where we will utilize an A-B-A, or return to baseline design where all participants will experience the intervention in between two baseline observation periods.
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Reinforcement, or incentives, in exchange for evidence of not drinking alcohol.

SUMMARY:
Alcohol abuse remains a significant cause of preventable morbidity and mortality in the US. Yet only 15% of those with alcohol use disorders receive treatment. Contingency Management (CM) is a cost-effective intervention for drug addiction where individuals are rewarded when they submit biological verification of drug abstinence. The researchers propose to develop an integrated CM system capable of incorporating mobile device input, that would allow them to deliver a CM intervention for problematic drinking to anyone who owns a smartphone. The mobile device input will incorporate ecological momentary assessments (EMA), geospatial mapping, and biomarker-based feedback from a portable measuring device.

DETAILED DESCRIPTION:
The researchers propose to develop an integrated Contingency Management (CM) system capable of incorporating mobile device input, which would allow them to deliver a CM intervention for problematic drinking to anyone who owns a smartphone. The location of participants through their cell phone will be recorded. The researchers will be using this data to create a "heat-map" to find problem areas of drinking. The application works only on iPhone 7 or a newer version with an (iPhone Operating System) iOS 13.5. If the participant does not have an iPhone 7 or a newer version, the researcher can loan one to the participant if he/she knows how to use it, but it must be returned at the end of the study.

The primary aim is to combine mobile technology, geospatial mapping, and biomarker measurement, with individual goal setting and ecological momentary assessments (EMA) feedback to launch behavioral modification strategies and progress monitoring.

People can participate if they are 1) age 18-65 years; 2) have an Alcohol Use Disorders Identification Test (AUDIT) score of 8 or higher; 3) have the ability to read and speak English; 4) have the ability to provide written informed consent; 5) have a breath alcohol of 0.00 during informed consent, and 6) can operate a smartphone with an active service provider.

The researchers will utilize an A-B-A completely within-subject design with the intent of recruiting twenty total participants from the Community in Spokane.

During the first A phase, participants will receive reinforcement for simply submitting breath samples 3 times per day between 4 and 6 hours apart.

During the B phase, the delivery of reinforcers will be contingent upon the submission of an alcohol negative breath sample on an escalating schedule.

The A phase or return to the baseline phase will involve the delivery reinforcers for simply submitting a sample during the designated windows of time.

The researchers will also collect other EMA data on stress, anxiety, depression, and other brief measures daily through participants' smartphone. Each phase will last a total of 4 weeks (i.e., 2 weeks of the first A phase, 4 weeks of the B phase, and then 2 more weeks of the A-phase) each for a total of 8 weeks of participation. Participants will be asked to submit 3 breath samples per day through a Bluetooth enabled breathalyzer developed by BACTrack no less than 8 hours apart and no more than 12 hours apart. Test results for breath alcohol will be available instantly to the participant and uploaded to the CM response system almost immediately.

As part of this CM system, participants will have the capability to receive multi-modal message reminders when they enter a new window of needed biochemical sample submission and additional reminders when the window of sample submission is about to close. While participants will receive information messages to this effect during the A phase, participants will receive additional personalized multi-modal message reminders once the CM platform can detect that they have entered a cold or hot zone. For example, upon entering a hot zone radius during the B phase wherein they had a greater 50% likelihood of drinking in that zone during the A phase, they will receive a text message encouraging them to change surroundings in order to better promote abstinence. Also, if the participant is within a window of time where they are eligible to submit a sample and receive a dose of reinforcement, this is another action that the individual can take to help bolster their attempt to remain abstinent. All these data (i.e., biochemical results, location of sample submission, time of submission, and other bits of data) will be collected and be presented in summary form to the research team. This will help the team devise an action plan if the participant's drinking behavior is proving impervious to intervention or if the participant's goals are being met, this is something the researcher can encourage about.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. An Alcohol Use Disorders Identification Test (AUDIT) score of 8 or higher.
3. Ability to read and speak English.
4. Ability to provide written informed consent.
5. Breath alcohol of 0.00 during informed consent.
6. Operate a smartphone with an active service provider.

Exclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) alcohol use disorder, severe type.
2. Significant risk of dangerous alcohol withdrawal, defined as a history of alcohol detoxification or seizure in the last 12 months and expression of concern by the participant about dangerous withdrawal.
3. Diagnosis of a psychotic disorder.
4. Lifetime suicide attempt or suicidality in the past year.
5. Any other medical or psychiatric condition that would compromise safe participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Contingency Management A-B-A
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Contingency Management A-B-A
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Employment [Count of Participants; unit: Participants]
  Employed | 9
  Unemployed | 3
Baseline EtG Result [Count of Participants; unit: Participants]
  Positive | 11
  Negative | 1

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Measured Change in Alcohol Abstinence.
Description: Change in biochemically measured alcohol abstinence assessed through breath samples submitted three times daily.
Time Frame: Daily during 8 weeks (2 weeks of first A phase, 4 weeks of B phase, and 2 second A phase)
Population: This is a within subject design (each participant goes through all three phases, the two A phases are control phases and B is the experimental phase). The overall number of units is total BAC submission for all phases. The numbers analyzed below differ based on total number of samples submitted by phase.
Measure: Number; unit: Number of negative BAC samples by phase.
Units Other Than Participants: Total BAC samples submitted
Arm/Group | Contingency Management A-B-A
Number analyzed (Participants) | 12
Number analyzed (Total BAC samples submitted) | 2016
Number of negative BAC samples by phase.
  First A Phase: number analyzed (Total BAC samples submitted) | 411
  First A Phase | 347
  B Phase: number analyzed (Total BAC samples submitted) | 700
  B Phase | 615
  Second A Phase: number analyzed (Total BAC samples submitted) | 249
  Second A Phase | 209

2. Secondary Outcome: Feasibility Indicator of App Usage
Description: Percentage of actual BAC samples submitted by the total number of possible submissions.
Time Frame: 8 weeks (2 weeks of first A phase, 4 weeks of B phase, and 2 second A phase)
Population: as for outcome 1
Measure: Number; unit: BAC samples actually submitted by phase
Units Other Than Participants: Total possible submissions of BAC sample
Arm/Group | Contingency Management A-B-A
Number analyzed (Participants) | 12
Number analyzed (Total possible submissions of BAC sample) | 2016
BAC samples actually submitted by phase
  First A Phase: number analyzed (Total possible submissions of BAC sample) | 504
  First A Phase | 411
  B Phase: number analyzed (Total possible submissions of BAC sample) | 1008
  B Phase | 700
  Second A Phase: number analyzed (Total possible submissions of BAC sample) | 504
  Second A Phase | 249

3. Secondary Outcome: Treatment Retention
Description: Duration in weeks of treatment retention
Time Frame: 8 Weeks
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Contingency Management A-B-A
Number analyzed (Participants) | 12
Weeks | 7.5 (1.1)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Description: Participants were asked once weekly at their visits about potential adverse events.
Groups:
- First A Phase: All participants will be assigned a single arm within subject design, where we will utilize an A-B-A, or return to baseline design where all participants will experience the intervention in between two baseline observation periods. Participants were asked weekly about adverse events over the course of 8 weeks.
  This arm reflects the 2 weeks in first A phase.
- B Phase: All participants will be assigned a single arm within subject design, where we will utilize an A-B-A, or return to baseline design where all participants will experience the intervention in between two baseline observation periods. Participants were asked weekly about adverse events over the course of 8 weeks.
  This arm reflects the 4 weeks in the experimental B phase.
- Second A Phase: All participants will be assigned a single arm within subject design, where we will utilize an A-B-A, or return to baseline design where all participants will experience the intervention in between two baseline observation periods. Participants were asked weekly about adverse events over the course of 8 weeks.
  This arm reflects the 2 weeks in the second A phase.
Arm/Group | First A Phase | B Phase | Second A Phase
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First A Phase (N=12) | B Phase (N=12) | Second A Phase (N=12)
Kidney Pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Related to over consumption of alcohol during first A phase. Participant 1.
Mild headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Mild headache believed to be due to wildfire smoke during first A phase. Participant 5.
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Sleep apnea believed to be due to smoking during B phase. Participant 1.
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Injury to shoulder, treated with ice during B Phase. Participant 11.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT04656925/Prot_000.pdf
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/25/NCT04656925/ICF_001.pdf